CLINICAL TRIAL: NCT05925699
Title: National Database of the Virtual Institute of Cerebrovascular Diseases
Acronym: BIG-MENTI
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Humanitas Hospital, Italy (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); I.R.C.C.S. Fondazione Santa Lucia (Other); Ospedale Policlinico San Martino (Other); IRCCS San Camillo, Venezia, Italy (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Ospedale Pediatrico Bambin Gesù (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); IRCCS Fondazione Stella Maris (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); IRCCS San Raffaele Roma (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Ospedale San Raffaele (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Istituto Auxologico Italiano (Other); Istituti Clinici Scientifici Maugeri SpA (Other); Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Principal Investigator, Calabresi Paolo, Professor, Head of Neurology Department, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5832
Record Dates: First submitted 2023-06-09; First posted 2023-06-29 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Cerebrovascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients with new-onset cerebrovascular disease from January 1, 2016 to July 1, 2049
  Interventions: Other: Collection of clinical, radiological, and biological data from patients' medical records

INTERVENTIONS:
Other: Collection of clinical, radiological, and biological data from patients' medical records — Collection of clinical, radiological, and biological data from patients' medical records

SUMMARY:
The primary aim of the study is to develop a national registry of cerebrovascular diseases in order to define the subtypes of these diseases associated with a worse prognosis. Secondly, the study aims to find clinical, radiological, and biological markers capable tof predicting the outcome of cerebrovascular diseases and the onset of complications related to therapeutic procedures, and to calculate predictive prognostic scores composed of multiple variables.

Each participating center will collect clinical, radiological, and biological data from the medical records of the study participants. Patients included in the study will not undergo any additional medical procedures to those of normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebrovascular pathology defined according to the NINDS special report of 1990 as "all disorders in which there is an area of the brain transiently or permanently affected by ischemia or bleeding and/or in which one or more blood vessels of the brain are mainly altered by a pathological process", falling within the following codes of the International Classification of Diseases, 9th revision (ICD-9): ICD-9 430-438;
* Informed consent provided by the patient or his legal representative in the case of mental incapacity or by the parents/guardians in the case of minors.

Exclusion Criteria:

* The patient, his legal representative in the case of mental incapacity or his parents/guardians in the case of minors clearly state their will to leave the study;
* Onset of cerebrovascular disease before January 1, 2016.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with cerebrovascular diseases occuring between January 1, 2016 and July 1, 2049 who consented to partecipate in the study
Sampling Method: Non-Probability Sample
Enrollment: 285600 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2052-09-01 (Estimated); Study Completion 2052-09-01 (Estimated)

PRIMARY OUTCOMES:
Identification of subtypes of each cerebrovascular disease (ICD-9 430-438) associated with poor prognosis. | July 1, 2023 - July 1, 2053
  Identification and definition of the various subtypes of each cerebrovascular disease (International Classification of Diseases, 9th revision (ICD-9): ICD-9 430-438) associated with poor prognosis.

SECONDARY OUTCOMES:
Identification of clinical variables of each cerebrovascular disease correlated with its prognosis | July 1, 2023 - July 1, 2053
  Identification of the clinical variables of each cerebrovascular disease correlated with its prognosis
Identification of radiological variables of each cerebrovascular disease correlated with its prognosis | July 1, 2023 - July 1, 2053
  Identification of the radiological variables of each cerebrovascular disease correlated with its prognosis
Identification of biomarkers of each cerebrovascular disease correlated with its prognosis | July 1, 2023 - July 1, 2053
  Identification of the biomarkers of each cerebrovascular disease correlated with its prognosis
Identification of neurophysiological variables of each cerebrovascular disease correlated with its prognosis | July 1, 2023 - July 1, 2053
  Identification of the neurophysiological variables of each cerebrovascular disease correlated with its prognosis
Identification of prognostic scores for each cerebrovascular disease | July 1, 2023 - July 1, 2053
  Identification of prognostic scores for each cerebrovascular disease, based on the combination of clinical, radiological, neurophysiological and biomarker variables
Identification of clinical variables of each cerebrovascular disease helping in differential diagnosis | July 1, 2023 - July 1, 2053
  Identification of clinical variables of each cerebrovascular disease that help the clinician in early differential diagnosis
Identification of clinical variables of each cerebrovascular disease capable of predicting the development of complications | July 1, 2023 - July 1, 2053
  Identification of clinical variables of each cerebrovascular disease capable of predicting the development of spontaneous complications or complications related to therapeutic procedures
Identification of clinical variables of each cerebrovascular disease able to predict the success of pharmacological or procedural therapies | July 1, 2023 - July 1, 2053
  Identification of clinical variables of each cerebrovascular disease able to predict the success of pharmacological or procedural therapies
Identification of the clinical variables of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome | July 1, 2023 - July 1, 2053
  Identification of the clinical variables of each cerebrovascular disease useful for the purpose of personalizing the rehabilitation treatment and able to predict the good functional outcome following the same rehabilitation treatments
Identification of neurophysiological variables of each cerebrovascular disease helping in differential diagnosis | July 1, 2023 - July 1, 2053
  Identification of neurophysiological variables and biomarkers of each cerebrovascular disease helping in differential diagnosis
Identification of radiological variables of each cerebrovascular disease helping in differential diagnosis | July 1, 2023 - July 1, 2053
  Identification of radiological variables of each cerebrovascular disease helping in differential diagnosis
Identification of neurophysiological variables of each cerebrovascular disease capable of predicting the development of complications | July 1, 2023 - July 1, 2053
  Identification of neurophysiological variables of each cerebrovascular disease capable of predicting the development of complications
Identification of radiological variables of each cerebrovascular disease capable of predicting the development of complications | July 1, 2023 - July 1, 2053
  Identification of radiological variables of each cerebrovascular disease capable of predicting the development of complications
Identification of biomarkers of each cerebrovascular disease helping in differential diagnosis | July 1, 2023 - July 1, 2053
  Identification of biomarkers of each cerebrovascular disease helping in differential diagnosis
Identification of biomarkers of each cerebrovascular disease capable of predicting the development of complications | July 1, 2023 - July 1, 2053
  dentification of biomarkers of each cerebrovascular disease capable of predicting the development of complications
Identification of biomarkers of each cerebrovascular disease able to predict the success of pharmacological or procedural therapies | July 1, 2023 - July 1, 2053
  Identification of biomarkers of each cerebrovascular disease able to predict the success of pharmacological or procedural therapies
Identification of radiological variables of each cerebrovascular disease able to predict the success of pharmacological or procedural therapies | July 1, 2023 - July 1, 2053
  Identification of radiological variables of each cerebrovascular disease able to predict the success of pharmacological or procedural therapies
Identification of the radiological variables of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome | July 1, 2023 - July 1, 2053
  Identification of the radiological variables of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome
Identification of the neurophysiological variables of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome | July 1, 2023 - July 1, 2053
  Identification of the neurophysiological variables of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome
Identification of the biomarkers of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome | July 1, 2023 - July 1, 2053
  Identification of the biomarkers of each cerebrovascular disease useful for the personalization of the rehabilitation treatment and able to predict its functional outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided
All the data collected in the registry will be available, upon reasonable request, for all the PIs and Sub-Is of the study of the various participating centers

REFERENCES:
- [Result] Special report from the National Institute of Neurological Disorders and Stroke. Classification of cerebrovascular diseases III. Stroke. 1990 Apr;21(4):637-76. doi: 10.1161/01.str.21.4.637. No abstract available. PMID 2326846
- [Result] Timmis A, Vardas P, Townsend N, Torbica A, Katus H, De Smedt D, Gale CP, Maggioni AP, Petersen SE, Huculeci R, Kazakiewicz D, de Benito Rubio V, Ignatiuk B, Raisi-Estabragh Z, Pawlak A, Karagiannidis E, Treskes R, Gaita D, Beltrame JF, McConnachie A, Bardinet I, Graham I, Flather M, Elliott P, Mossialos EA, Weidinger F, Achenbach S; Atlas Writing Group, European Society of Cardiology. European Society of Cardiology: cardiovascular disease statistics 2021. Eur Heart J. 2022 Feb 22;43(8):716-799. doi: 10.1093/eurheartj/ehab892. PMID 35016208
- [Result] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Result] Sacco S, Stracci F, Cerone D, Ricci S, Carolei A. Epidemiology of stroke in Italy. Int J Stroke. 2011 Jun;6(3):219-27. doi: 10.1111/j.1747-4949.2011.00594.x. PMID 21557809
- [Result] Ozpinar A, Mendez G, Abla AA. Epidemiology, genetics, pathophysiology, and prognostic classifications of cerebral arteriovenous malformations. Handb Clin Neurol. 2017;143:5-13. doi: 10.1016/B978-0-444-63640-9.00001-1. PMID 28552158
- [Result] Ferro JM, Aguiar de Sousa D. Cerebral Venous Thrombosis: an Update. Curr Neurol Neurosci Rep. 2019 Aug 23;19(10):74. doi: 10.1007/s11910-019-0988-x. PMID 31440838

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05925699/Prot_SAP_000.pdf